CLINICAL TRIAL: NCT03726437
Title: RealConsent: A Web-based Program to Reduce College Women's Risk of Sexual Violence by Targeting Alcohol Use, Communication and Consent, and Building Supportive Networks
Brief Title: Efficacy of a Web-based Sexual Violence Risk Reduction Program for Female College Students
Acronym: RealConsent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Behavioral Science Technologies, LLC (Industry)
Responsible Party: Principal Investigator, Laura F Salazar, Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R42AA025817-03 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sexual Violence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were told that study was to determine efficacy of a web-based health promotion program for female freshmen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RealConsent (Experimental): A 3-hour web-based program designed to teach female college freshmen strategies to reduce their risk of sexual violence victimization.
  Interventions: Behavioral: RealConsent
- Stress and Mood Management (Placebo Comparator): A 3-hour general mental health web-based program.
  Interventions: Behavioral: Stress and Mood Management

INTERVENTIONS:
Behavioral: RealConsent — This 3-hour web-based program consists of four 45-minute modules that are interactive and range in number of segments (1-14) and types of activities. Each of the modules involves interactivity, didactic activities and two episodes of a serial drama ("Squad"), which allow for the modeling of positive behaviors and illustrate both positive and negative outcome expectations. Behaviors modeled include drinking safely (e.g., eating before drinking, pacing, and drinking water), having a game plan before going out, communicating with male sex partners, engaging in protective dating behaviors, use of resistance strategies, self-defense strategies and bystander intervention with the goal of reducing risk of being sexually assaulted.
  Arms: RealConsent
Behavioral: Stress and Mood Management — This 3-hour general health promotion web-based program consists of four 45-minute modules ("Stress Management", "Managing Depression", "Managing Anxiety", and "Treatments that work") that provide a range of activities related to reducing day-to day stress and alleviating anxiety through meditation and exercise.
  Arms: Stress and Mood Management

SUMMARY:
This study evaluates the efficacy of a web-based program for female college freshmen ("RealConsent") in reducing their risk of sexual violence victimization. Half the participants will receive RealConsent-F and half will receive an attention-placebo control ("Stress and Mood Management").

DETAILED DESCRIPTION:
Sexual assault of college women is a serious and complex public health problem: one in five college women report being sexually assaulted. The purpose of this study is to conduct a randomized controlled trial study with 750 female college students from three universities to test the efficacy of RealConsent, a sexual violence risk reduction program for college women, compared to an attention-placebo control. RealConsent is a multi-media 3-hour program based on social cognitive theory and alcohol myopia theory. The primary outcome will be self-reported sexual violence victimization and the secondary outcomes will be alcohol and dating protective- and risk-related behaviors and resistance strategies. The investigators expect that women in the treatment group will report less sexual violence victimization than women in the control group. Expected outcomes are demonstrated feasibility and efficacy of a technologically novel risk reduction program for female college students.

ELIGIBILITY:
Inclusion Criteria:

* female, aged 18-20 years, full-time freshmen, matriculated at Georgia State University, Emory University, or University of Georgia, and single (i.e., not in a committed dating relationship).

Exclusion Criteria:

* other education levels, married, and/or graduate status

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 881 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura F. Salazar, PhD, Principal Investigator — Georgia State University; Anne Marie Schipani-McLaughlin, PhD, Study Director — Georgia State University; George Cavagnaro, MBA, Study Chair — Behavioral Science Technologies, LLC
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from approximately 750 female freshmen participating in this study will be made available. The final dataset will include self-reported sexual violence victimization experiences, risk behaviors and scale measures of secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: The study principal investigator will review all data requests. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Salazar LF, Schipani-McLaughlin AM, Sebeh Y, Nizam Z, Hayat M. A Web-Based Sexual Violence, Alcohol Misuse, and Bystander Intervention Program for College Women (RealConsent): Randomized Controlled Trial. J Med Internet Res. 2023 Jun 21;25:e43740. doi: 10.2196/43740. PMID 37342080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RealConsent | Stress and Mood Management
Started (Randomized to RealConsent) | 444 | 437 (Randomized to Attention placebo group)
Completed (Completed 6-month follow-up assessments.) | 359 | 361 (Completed 6-month follow-up assessment)
Not Completed | 85 | 76
Not completed — Lost to Follow-up | 85 | 76

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RealConsent | Stress and Mood Management | Total
Number analyzed (Participants) | 444 | 437 | 881
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 444 | 437 | 881
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 437 | 881
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 91 | 90 | 181
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 103 | 110 | 213
  White | 198 | 196 | 394
  More than one race | 47 | 37 | 84
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 444 | 437 | 881
Sexual Violence Victimization [Mean (Standard Deviation); unit: scores on a scale] — Sexual assault victimization was assessed with Revised Sexual Experiences Survey. Participants were asked how often they experienced 7 unwanted sexual experiences. Also, the tactic that was used ("using force") was also noted. Response options ranged from 0 (never) to 3 (3+times). An overall score for the SES, was calculated by summing each outcome and tactic score ("SOTS") with a range from 0 to 135- with higher scores indicating more sexual violence victimization. The 2nd method combines several of the outcomes, but keeps tactics separate, resulting in a potential range of 0 to 63.
  scores on a scale
    Sexual Violence Vict. "SOTS" | 5.6 (15.7) | 5.7 (17.1) | 5.7 (16.4)
    Sexual Violence Vict. "COSTS" | 3.7 (8.9) | 3.8 (9.8) | 3.7 (9.4)
Alcohol Protective Behaviors [Mean (Standard Deviation); unit: scores on a scale] — Alcohol protective behaviors was measured by a scale developed by Martens et al., 2005 that included 15 protective strategies (e.g.., "alternate alcoholic and non-alcoholic drinks") that asked participants if they had engaged in within the last 3 months. with response options of Never (1) to Always (5). Responses were summed across the 15 items. Potential range was 15 to 75. Higher scores indicated MORE protective strategies were used.
  scores on a scale | 53.53 (12.2) | 53.97 (11.4) | 53.76 (11.76)
Dating Risk Behaviors [Mean (Standard Deviation); unit: scores on a scale] — Dating Risk Behaviors were measured by the Dating Behavior Survey created by Hanson & Gidycz, 1993. The scale consists of 15 items that assess different situational variables (e.g., "consuming alcohol on the first date") that have been found to be related to sexual violence victimization. Participants are asked to respond how often they have engaged in the behavior on the first few dates with a new partner. Response options ranged from Never (1) to Always (5). Scores are summed and higher scores indicate engaging in MORE risk behaviors. Overall scores can range from 15 to 75.
  scores on a scale | 35.16 (5.1) | 35.08 (4.8) | 35.12 (4.96)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sexual Violence Victimization at 6-months Follow-up
Description: Sexual assault victimization was assessed with Revised Sexual Experience Survey. Participants were asked how often they experienced 7 unwanted sexual experiences. Also, the tactic that was used ("using force") was also noted. Response options ranged from 0 (never) to 3 (3+times). An overall score for the SES, was calculated by summing each outcome and tactic score ("SOTS") with a range from 0 to 135- with higher scores indicating more sexual violence victimization. The 2nd method combines several of the outcomes, but keeps tactics separate, resulting in a potential range of 0 to 63.
Time Frame: Baseline to 6-months
Population: Intent-to-treat population (all RealConsent and Stress and Mood Management participants from whom we had data at 6-month follow-up).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 359 | 361
score on a scale
  Baseline score of "SOTS" | 5.64 (15.67) | 5.68 (17.10)
  6-Month score of "SOTS" | 5.52 (18.4) | 8.15 (25.36)
  Baseline score of "COSTS" | 3.69 (8.93) | 3.78 (9.77)
  6-Month score of "COSTS" | 3.52 (10.55) | 4.95 (13.63)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority — Analyses were performed to determine whether RealConsent was superior to Stress and Mood Management in reducing incidence of sexual violence victimization; p = .0002, Mixed Models Analysis; Models adjusted for fixed effects; Risk Ratio (RR) = .48, 95% CI 2-sided [.33 to .69]
Statistical Analysis 2: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p = .31, Mixed Models Analysis; Models adjusted for fixed effects; Odds Ratio (OR) = .77, 95% CI 2-sided [.47 to 1.28]

2. Secondary Outcome: Change From Baseline in Alcohol Protective Behaviors at 6 Months
Description: Alcohol protective behaviors was measured by a scale developed by Martens et al., 2005 that included 15 protective strategies (e.g.., "alternate alcoholic and non-alcoholic drinks") that asked participants if they had engaged in within the last 3 months. with response options of Never (1) to Always (5). Responses were summed across the 15 items. Potential range was 15 to 75. Higher scores indicated MORE protective strategies were used.
Time Frame: Baseline to 6 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 359 | 361
score on a scale
  Baseline | 53.53 (12.17) | 53.97 (11.35)
  6 months | 56.8 (11.7) | 55.0 (11.6)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p = .03, Mixed Models Analysis; Model adjusted for fixed effects; Adjusted OR = 1.17, 95% CI 2-sided [0.12 to 1.22]

3. Secondary Outcome: Change From Baseline in Dating Risk Behaviors at 6-months Follow-up
Description: Dating Risk Behaviors were measured by the Dating Behavior Survey created by Hanson & Gidycz, 1993. The scale consists of 15 items that assess different situational variables (e.g., "consuming alcohol on the first date") that have been found to be related to sexual violence victimization. Participants are asked to respond how often they have engaged in the behavior on the first few dates with a new partner. Response options ranged from Never (1) to Always (5). Scores are summed and higher scores indicate engaging in MORE risk behaviors. Overall scores can range from 15 to 75.
Time Frame: Baseline to 6 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 359 | 361
score on a scale
  Baseline | 35.16 (5.11) | 35.08 (4.80)
  6 months | 36.2 (7.3) | 36.1 (5.7)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p < .05, Mixed Models Analysis; Model adjusted for fixed effects; Adjusted OR = -.50, 95% CI 2-sided [-1.27 to 0.27]

4. Secondary Outcome: Change From Baseline in "Number of Times Engaged in Binge Drinking" to 6-months
Description: Participants were asked at baseline and at 6-month follow-up, to report: "In the past 30 days, the number of times four or more drinks were consumed in one setting."
Time Frame: Baseline to 6-months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Binge drinking events
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 359 | 361
Binge drinking events
  Baseline | 1.71 (2.53) | 1.25 (1.8)
  6 months | 1.11 (1.8) | 1.05 (1.8)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p = .02, Mixed Models Analysis; Model adjusted for fixed effects; Incidence rate ratio = .81, 95% CI 2-sided [.67 to .97]

5. Secondary Outcome: Change From Baseline in "Average Number of Alcoholic Drinks Per Occasion in Last 30 Days" to 6-months
Description: Participants were asked at baseline and at 6-month follow-up to report, "the average number of alcoholic drinks consumed per occasion in the last 30 days."
Time Frame: baseline to 6-months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Average number of drinks/occasion
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 359 | 361
Average number of drinks/occasion
  Baseline | 1.64 (1.3) | 1.45 (1.12)
  6 Months | 1.4 (1.2) | 1.3 (1.3)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p = .43, Mixed Models Analysis; Model adjusted for fixed effects; Incidence rate ratio = 1.05, 95% CI 2-sided [.92 to 1.20]

6. Secondary Outcome: Change From Baseline in Bystander Behavior at 6-months
Description: Bystander behavior was assessed using the 20-item Bystander Behavior Scale. Items assessed whether participants engaged in bystander behaviors in the past three months and included items such as, "If I saw someone taking a very intoxicated person up to their room, I said something and asked what the friend was doing." Higher scores indicate a better outcome of engaging in more prosocial behaviors. Min value=0; Max value=60.
Time Frame: Baseline to 6-months
Population: Analysis was performed using dosage were: (1) the RealConsent® group participants at 6-months who completed all four modules (n=305) versus the RealConsent® group participants who had not completed all four modules plus the control group participants (n=415).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RealConsent | Stress and Mood Management
Number analyzed (Participants) | 305 | 415
score on a scale
  Baseline | 7.14 (9.02) | 6.58 (9.03)
  6 Months | 6.03 (8.1) | 7.6 (11.14)
Statistical Analysis 1: Comparison: RealConsent vs Stress and Mood Management; Test type: Superiority; p = .006, Mixed Models Analysis; Model adjusted for fixed effects; Adjusted OR = 1.72, 95% CI 2-sided [1.17 to 2.55]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | RealConsent | Stress and Mood Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03726437/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03726437/ICF_000.pdf